CLINICAL TRIAL: NCT05419011
Title: A Phase IIB Clinical Trial of the Multitargeted Recombinant Adenovirus 5 (CEA/MUC1/Brachyury) Vaccines (TRI-AD5) and IL-15 Superagonist N-803 in Lynch Syndrome
Brief Title: Testing a Combination of Vaccines for Cancer Prevention in Lynch Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2021-14234; NCI-2021-14234 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI 21-05-01; NCI21-05-01 (Other: Northwestern University); INT21-05-01 (Other: DCP); P30CA060553 (NIH); UG1CA242596 (NIH); UG1CA242609 (NIH); UG1CA242632 (NIH); UG1CA242635 (NIH); UG1CA242643 (NIH)
Record Dates: First submitted 2022-06-14; First posted 2022-06-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Carcinoma; Colorectal Neoplasm; Lynch Syndrome
MeSH Terms: conditions — Colorectal Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Biopsy; Specimen Handling; Colonoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm I (Tri-Ad5, N-803) (Experimental): Participants receive Tri-Ad5 SC and N-803 SC at weeks 0, 4, 8, and 52. Participants also undergo SOC colonoscopy with biopsy at baseline and at 52 and 104 weeks. Participants undergo blood sample collection throughout the study.
  Interventions: Biological: Adenovirus 5 CEA/MUC1/Brachyury Vaccine Tri-Ad5; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Colonoscopy; Drug: Nogapendekin Alfa; Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): Participants receive placebo SC at weeks 0, 4, 8, and 52. Participants also undergo SOC colonoscopy with biopsy at baseline and at 52 and 104 weeks. Participants undergo blood sample collection throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Colonoscopy; Drug: Placebo Administration; Other: Questionnaire Administration
- Safety phase I (Tri-Ad5) (Experimental): Participants receive Tri-Ad5 SC at weeks 0, 4, 8, and 52. Participants also undergo SOC colonoscopy with biopsy at baseline and at 52 weeks and 104 weeks. Participants undergo blood sample collection throughout the study.
  Interventions: Biological: Adenovirus 5 CEA/MUC1/Brachyury Vaccine Tri-Ad5; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Colonoscopy; Other: Questionnaire Administration
- Safety phase II (Tri-Ad5 , N-803) (Experimental): Participants receive Tri-Ad5 SC and N-803 SC at weeks 0, 4, 8, and 52. Participants also undergo SOC colonoscopy with biopsy at baseline and at 52 weeks and 104 weeks. Participants undergo blood sample collection throughout the study.
  Interventions: Biological: Adenovirus 5 CEA/MUC1/Brachyury Vaccine Tri-Ad5; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Colonoscopy; Drug: Nogapendekin Alfa; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Adenovirus 5 CEA/MUC1/Brachyury Vaccine Tri-Ad5 — Given SC
  Other Names: Ad5 CEA/MUC1/Brachyury Vaccine Tri-Ad5; Ad5-CEA/Ad5-MUC1/Ad5-Brachyury Vaccine Tri-Ad5; Adenoviral CEA/MUC1/Brachyury Vaccine Tri-Ad5; Tri Ad5; Tri-Ad5; TriAd5
  Arms: Arm I (Tri-Ad5, N-803); Safety phase I (Tri-Ad5); Safety phase II (Tri-Ad5 , N-803)
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Colonoscopy — Undergo SOC colonoscopy
Drug: Nogapendekin Alfa — Given nogapendekin alfa inbakicept (N-803) SC
  Arms: Arm I (Tri-Ad5, N-803); Safety phase II (Tri-Ad5 , N-803)
Drug: Placebo Administration — Given SC
  Arms: Arm II (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase IIb trial tests whether Tri-Ad5 in combination with N-803 works to prevent colon and other cancers in participants with Lynch syndrome. Each of the three injections in Tri-Ad5 vaccine contain a different substance that is in precancer and cancer cells. Injecting these substances may cause the immune system to develop a defense against cancer that recognizes and destroys any precancer and cancer cells that produce these proteins in the future. N-803 may increase immune responses to other vaccines. Giving Tri-Ad5 in combination with immune enhancing N-803 may lower the chance of developing colon and other cancers in participants with Lynch syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate if the combination of trivalent adenovirus-5 (Tri-Ad5) vaccines and IL-15 superagonist nogapendekin alfa inbakicept (N-803) reduces the incidence of colorectal neoplasms in patients with Lynch syndrome (LS).

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of the Tri-Ad5 vaccines + N-803 in combination.

II. To correlate clinical factors such as use of aspirin and non-steroidal anti-inflammatory drugs (NSAID), smoking and alcohol intake with immune responses.

III. To evaluate the effect of Tri-Ad5 vaccines on the incidence of LS-related extracolonic cancers.

IV. To systematically measure the participants' behavior and experience in terms of vaccine uptake, cancer-specific distress and quality of life.

EXPLORATORY OBJECTIVES:

I. To determine the ability of the Tri-Ad5 vaccines + N-803 to generate a 2-fold increase in T cell responses (cell-mediated immunity) at week 12 (early immune response) and at week 56 (long-term memory response).

II. To evaluate circulating anti-MUC1 IgG (antibody-mediated immunity) after Tri-Ad5 vaccines + N-803.

III. To compare the expression of the three tumor associated antigen (TAAs): MUC1, carcinoembryonic antigen (CEA) and brachyury in colorectal neoplasms before and after Tri-Ad5 vaccines + N-803.

IV. To evaluate changes in the immune profile and abundance of resident immune cell types in colonic mucosa after vaccination with Tri-Ad5 vaccines + N-803 using messenger ribonucleic acid sequencing (mRNAseq) and immunohistochemistry (IHC).

V. To test the effects of the vaccines alone or in combination with N-803 on specific immune subsets of peripheral blood mononuclear cells (PBMCs) and serum soluble factors and cytokines.

VI. To compare the expression of stem cell markers in colorectal neoplasms before and after Tri-Ad5 vaccines + N-803.

VII. To compare the number of mismatch repair deficient (MMR-deficient) crypts at baseline to the number of MMR-deficient crypts at the one year post-vaccination colonoscopy both overall and on a per patient basis.

OUTLINE:

SAFETY PHASE I: Participants receive Tri-Ad5 subcutaneously (SC) at weeks 0, 4, 8, and 52. Participants also undergo standard of care (SOC) colonoscopy with biopsy at baseline, at 52 weeks and 104 weeks.

SAFETY PHASE II: Participants receive Tri-Ad5 SC and N-803 SC at weeks 0, 4, 8, and 52. Participants also undergo SOC colonoscopy with biopsy at baseline, 52 weeks and 104 weeks.

RANDOMIZED CONTROL PHASE: Participants are randomized into 1 of two arms.

ARM I: Participants receive Tri-Ad5 SC and N-803 SC at weeks 0, 4, 8, and 52. Participants also undergo SOC colonoscopy with biopsy at baseline and at 52 and 104 weeks.

ARM II: Participants receive placebo SC at weeks 0, 4, 8, and 52. Participants also undergo SOC colonoscopy with biopsy at baseline and at 52 and 104 weeks.

Participants undergo blood sample collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with LS defined as one of the following:

  * Mutation positive: MLH1, MSH2/EPCAM and MSH6 genotypes with prior history of ≥1 colorectal neoplasms** (tubular or tubulovillous adenoma[s] or sessile serrated polyps/adenomas/lesion[s] or traditional serrated adenoma[s]), and/or colorectal cancer[s] (but no active cancer for 6 months) OR
  * PMS2 genotype with prior history of colon cancer(s) (but no active cancer for 6 months)

    * Note: Should be confirmed by pathology report or letter from endoscopist to participant
* Participants must have at least part of the descending/sigmoid colon and/or rectum intact
* Participants must be at least 6 months from any cancer-directed treatment (such as surgical resection, chemotherapy, immunotherapy or radiation). Ongoing adjuvant endocrine therapy is allowed
* Participants >= 18 years will be enrolled. Because the risk of LS related cancers is very low in participants < 18 years of age, children and adolescents are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Platelets >= 100,000/microliter
* Total bilirubin =< institutional upper limit of normal

  * Note: Higher bilirubin levels (<= 3 mg/dL) can be allowed if due to a known benign liver condition, i.e. Gilbert's
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional upper limit of normal
* Creatinine =< institutional upper limit of normal or estimated glomerular filtration rate (eGFR) >= 60 ml/min/1.73m^2
* The effects of the Tri-Ad5 vaccines and N-803 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Participants must be willing and able to space coronavirus disease (COVID) vaccines at least 2 weeks prior to and 2 weeks after receipt of study agent

Exclusion Criteria:

* History of organ allograft or other history of immunodeficiency
* Known human immunodeficiency virus (HIV) with CD4 count < 540, hepatitis B virus (HBV), or hepatitis C virus (HCV) infection. Subjects with laboratory evidence of cleared HBV and HCV infection will be permitted. Poorly controlled HIV may prevent an adequate immune response to the vaccine and will be an exclusion criterion
* Subjects requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 3 months of vaccination
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to adenovirus-based vaccines and N-803
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because of the unknown effects of the vaccine and N-803 on the fetus. Because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with the vaccine plus N-803, breastfeeding should be discontinued if the mother is treated with the vaccine plus N-803
* History of untreated thrombotic disorders
* Participants who experienced severe side effects or allergic reactions to previous adenovirus-based vaccines (such as Johnson and Johnson COVID vaccine) will be excluded
* History of atrial fibrillation
* History of gastrointestinal hemorrhage and intracranial hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence rate of the composite endpoint of adenomas (tubular, tubulovillous and serrated), advanced adenomas and colon cancer | At 104 weeks
  Will be compared between the two arms using a stratified Cochran-Mantel-Haenszel test where the randomization stratification factors will be included as strata. The cumulative events rates will be reported for each study arm along with the corresponding two-sided 95% confidence intervals.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 104 weeks
  Identify the adverse events using Common Terminology Criteria for Adverse Events version 5.0.
Association of clinical factors with immune responses | At 104 weeks
  Will be evaluated by conducting univariate and multivariate binary regression analyses. These analyses will be conducted for both arms combined (in which case arm is included as a stratification factor in the model) and each arm separately. The proportions of cells within adenomas expressing stem cells markers pre- and post-vaccination will be compared within each study arm using the signed rank test, and within-subject changes will be compared between responders and non-responders using Wilcoxon rank-sum test for each arm separately and both arms combined. Comparisons between study arms will be conducted using a Wilcoxon rank-sum test.
Incidence of extracolonic neoplasms | At 104 weeks
  Will compare the observed incidences of lynch syndrome (LS)-related extracolonic cancers to historical control incidence of LS-related extracolonic cancers in this patient population. We will collect the information about extracolonic cancers by asking the participants and by reviewing the pathology reports for confirmation.
Participants' behavior and experience | At baseline, 12 weeks and 52 weeks
  Descriptive statistics will be used to summarize the results.

OTHER OUTCOMES:
Tumor antigen specific T cell responses (cell-mediated immunity) | At weeks 0, 4, 8, and 12
  Will be log-transformed before conducting any analyses. Comparisons of number of antigen-specific T-cells, PBMCs, serum soluble factors and antibodies between study arms will be conducted using a nonparametric Wilcoxon rank sum test. IgG titers that will be measured serially will be analyzed and compared between the two arms using linear mixed effects models. If zero-inflation is detected, generalized linear mixed models with zero-inflated Poisson or negative binomial distributions will be fitted.
Circulating anti-MUC1 IgG (antibody-mediated immunity) | At baseline, 52 weeks, and 104 weeks
  Will be reported using repeated measures techniques. We will also compare pre- and post-vaccination size, number and histology of polyps.
Differential expression analyses | At baseline, 52 weeks, and 104 weeks
  Will be using Bioconductor R package DESeq2. A paired sample design to compare post- to pre-vaccination samples within each study arm and for both arms combined. Significant genes with Benjamini-Hochberg-adjusted p-value =< 0.05 and absolute value of log2-fold change >= 0.5 will be annotated with pathways of interest in volcano plots.
Immune cell gene enrichment analysis | At baseline, 52 weeks, and 104 weeks
  Will be calculated using raw read counts with Bioconductor R package GSVA.
Immune subsets of peripheral blood mononuclear cell and serum soluble factors and cytokine | At baseline, 52 weeks, and 104 weeks
  Will be calculated using raw read counts with Bioconductor R package GSVA.
Expression of stem cell markers | At baseline, 52 weeks, and 104 weeks
  Will be calculated using raw read counts with Bioconductor R package GSVA.
Number of mismatch repair deficient (MMR)-deficient crypts | At baseline and 1 year post-vaccination colonoscopy
  Will compare both overall and on a per patient basis. For patients with germline MMR variants and a known cancer history, MMR immunohistochemistry (IHC) will be performed based on the abnormal results in the patient's carcinoma and the germline MMR variant identified. For Lynch syndrome patients with no cancer history, IHC will be performed based on the affected MMR gene. Loss of MMR expression in non-neoplastic colonic crypts will be defined as complete absence of nuclear staining within the crypt epithelial cells within the crypt bases with concurrent nuclear expression in adjacent neighboring crypts, stromal cells, and lymphocytes. The number of crypt bases with loss of protein expression, if any, will be recorded. MMR protein-deficient non-neoplastic crypts will be further categorized based on the number of crypts exhibiting loss of protein expression. Single, isolated crypts with loss of MMR protein expression will be classified as solitary.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Bansal, Principal Investigator — University of Kansas
Locations (14):
- United States (13):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - University of Arizona Cancer Center - Prevention Research Clinic, Tucson, Arizona
  - UCSF Medical Center-Parnassus, San Francisco, California
  - University of Colorado, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
- University of Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
'NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page'
URL: https://grants.nih.gov/policy/sharing.htm